CLINICAL TRIAL: NCT05146921
Title: Gut Health and Probiotics in Parkinson's (SymPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KCH19-085
Record Dates: First submitted 2021-11-02; First posted 2021-12-07 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- food supplement: multi-strain probiotic (Symprove) (Active Comparator): 70 ml daily for 12 weeks
  Interventions: Dietary Supplement: Multi-strain probiotic
- Placebo (Placebo Comparator): 70 ml daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotic — The intervention in this study is a multi-strain probiotic which contains four live strains of bacteria:
  Lacticaseibacillus rhamnosus NCIMB 30174 Enterococcus faecium NCIMB 30176 Lactobacillus acidophilus NCIMB 30175 Lactiplantibacillus plantarum NCIMB 30173
  10 billion colony-forming units (CFU) per 70 ml cup
  Other Names: Symprove
  Arms: food supplement: multi-strain probiotic (Symprove)
Other: Placebo — placebo similar in appearance and taste to the active intervention but with no active bacteria
  Arms: Placebo

SUMMARY:
Current literature suggests that the gut microbiota is altered in patients with Parkinson's disease (PD) and might play a role in the clinical presentation and pathogenesis of this condition. The latter has driven the interest in investigating the use of gut microbiota-modulating interventions, such as probiotics, as possible novel therapeutic strategies for PD. Symprove is a food supplement working as an oral active probiotic which unlike many commercially available probiotics can reach the intestine and has been shown to be beneficial for gut health in gastrointestinal disorders.To date, no research has explored the possible effects of the intake of Symprove in PD. This is an exploratory study with a randomised, double-blind, placebo-controlled design investigating the effects of a 12-week probiotic intervention (Symprove) on gut and general health in 60 patients with PD and constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and upwards
* Diagnosis of idiopathic Parkinson's disease according to the Movement Disorder Society clinical diagnostic criteria
* Hoehn Yarh stage II-IV
* Diagnosis of constipation according to the ROME IV criteria and ≤ than 3 complete bowel movements per week

Exclusion Criteria:

* Diagnosis or suspicion of other causes for parkinsonism
* Advanced-stage therapies (deep brain stimulation, intrajejunal levodopa infusion, and apomorphine subcutaneous infusion)
* Any inflammatory bowel disease or diseases of the colon
* Previous surgery on the gastrointestinal tract
* History of laxative abuse
* Ongoing artificial nutrition
* Regular use of probiotics
* Previous intolerance and/or adverse reactions to probiotics
* Previous use of Symprove
* Recent or current use of any antibiotics (within 4 weeks before the start of the study)
* Swallowing issues interfering with the safety intake of the probiotic/placebo
* Pregnancy or lactation
* Major systemic disease
* Any condition interfering with the ability to give the informed consent
* Enrolment in another simultaneous investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota of study population | Baseline
  Gut microbiota will be evaluated with shallow shotgun sequencing of stool samples
Changes of gut microbiota following probiotic intervention and their association with changes in Parkinson's symptoms | 12 weeks
  Gut microbiota changes will be evaluated with shallow shotgun sequencing of stool samples while Parkinson's symptoms changes will be evaluated with subjective and objective measurements

SECONDARY OUTCOMES:
Blood | 12 weeks
  Changes in blood levels of inflammatory markers (i.e. C-reactive protein, cytokines, tight junction proteins, and short-chain fatty acids levels)

CONTACTS AND LOCATIONS:
Overall Officials: K Ray Chaudhuri, Professor, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom